CLINICAL TRIAL: NCT06579807
Title: Effect of a Cardiovascular Rehabilitation Program on Atherosclerosis, Endothelial Function and Inflammation in Patients With Coronary Artery Disease
Brief Title: Cardiac Rehabilitation and Coronary Artery Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia de Laranjeiras (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Juliana Pereira Borges, Principal investigator, Rio de Janeiro State University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 404204/2023-6
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Cardiac rehabilitation; Physical training; Inflammation; Intercellular adhesion molecules
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Inflammation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise training (Experimental): The multimodal supervised exercise program will include aerobic, resistance, and flexibility exercises during 12 weeks, performed in 3 weekly sessions lasting 60 minutes each.
  Interventions: Behavioral: Exercise training
- Control healthy (No Intervention): A reference group composed of healthy individuals without intervention will be included.

INTERVENTIONS:
Behavioral: Exercise training — The multimodal supervised exercise program will include aerobic, resistance, and flexibility exercises. The training program will last 12 weeks, performed in 3 weekly sessions lasting 60 minutes each. Aerobic exercise, lasting between 20-30 minutes, will be conducted on a treadmill or stationary bike at an intensity ranging from 75-85% of the maximal heart rate (HR), based on the cardiopulmonary exercise testing. Resistance training, lasting 30 minutes, will include 8 to 10 exercises performed in 3 sets of 10 to 12 maximum repetitions with 1-minute intervals, targeting major muscle groups of the upper and lower limbs, with loads corresponding to 80-90% of the 10-repetitions maximum (RM).
  Arms: Exercise training

SUMMARY:
Patients with coronary artery disease (CAD) aged 40-70 years will undergo exercise training (thrice weekly for 12 weeks). A reference group composed of healthy individuals will be included. Evaluations will be conducted at baseline and after the intervention period during two visits. During the first visit, carotid artery thickness will be assessed via ultrasound before and after a cardiopulmonary exercise testing. The second visit will include the evaluation of endothelial function using venous occlusion plethysmography. After this, participants will engage in 30 minutes of moderate-intensity aerobic exercise, and blood samples will be collected pre- and post-exercise. Circulating levels of kynurenine pathway (KP) metabolites (Tryptophan, kynurenine, kynurenic acid, and quinolinic acid), pro-inflammatory cytokines, cell adhesion molecules, and lipid profiles will be measured via Enzyme-Linked Immunosorbent Assay (ELISA), multiplex essays, and biochemical analysis; respectively.

DETAILED DESCRIPTION:
Participants and recruitment: In this clinical trial, 28 patients with CAD will be enrolled from the Pedro Ernesto University Hospital (HUPE) and 22 control volunteers without evidence of CAD (CTL) will be randomly recruited from among employees and students at the University of Rio de Janeiro State (UERJ). The groups will be matched by age and habitual physical activity level, assessed by the Baecke questionnaire, which quantifies activities performed at home, work, and leisure (sports).

All participants will receive oral and written instructions regarding the risks and benefits of the study and will provide written informed consent. The study was approved by the Research Ethics Committee of HUPE (CAAE 81718324.3.0000.5259). The study also adheres to SPIRIT 2013 (Standard Protocol Items: Recommendations for International Trials).

Study design: Evaluations will be conducted at baseline and after the 12-week intervention period during two visits interspersed by at least 72-hours interval. Outcomes in the CTL group will be assessed only at baseline to provide reference values. Visits will take place at the Physical Activity and Health Promotion Laboratory (LABSAU) and the Clinical and Experimental Research Laboratory on Vascular Biology (BioVasc), always in the morning (8:00 - 11:00 am), in rooms with controlled temperatures between 22°-24°C and relative humidity between 60-70%. Participants will be instructed to avoid physical activity, alcohol, and stimulants 48 hours prior to assessments.

During the first visit, volunteers will undergo a medical history assessment. If eligible, they will read and sign the informed consent form, if they agree to participate. Subsequently, carotid intima-media thickness will be assessed via carotid ultrasound, followed by a cardiopulmonary exercise testing (CPET). Immediately after the test, carotid intima-media thickness will be reassessed.

On the second visit, patients will undergo blood collection after 8 hours of fasting, followed by an assessment of vascular function using venous occlusion plethysmography. Approximately 15 min after a light standardized breakfast, participants will engage in 30 minutes of moderate-intensity aerobic exercise, after which blood samples will be collected again.

ELIGIBILITY:
Inclusion Criteria:

* Eligible CAD patients will be those aged 40 to 70 years, of both sexes, entering the cardiac rehabilitation program at HUPE. CAD will be defined as any acute coronary syndrome, including myocardial infarction with and without ST-segment elevation, and unstable angina (all defined by characteristic histories, electrocardiographic abnormalities, and cardiac enzyme abnormalities), or obstructive CAD diagnosed via coronary angiography (defined as ≥ 50% stenosis of any epicardial coronary artery) in patients with stable angina.
* Healthy controls: adults aged 40 to 70 years, of both sexes, without CAD evidence.

Exclusion Criteria:

* diagnosis of heart failure, pulmonary disease, Chagas disease, or tuberculosis
* regular physical exercise practice (≥ 3 days/week for 30 min) over the past 6 months
* malnutrition (body mass index [BMI] < 18.5 kg/m²)
* smoking
* obesity (BMI ≥ 30 kg/m²)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Carotid intima-media thickness | Baseline and 12 weeks
  The assessment of the intima-media thickness (IMT) of the left and right common carotid arteries will be performed with the patient in the supine position, with the head turned to the side (45°), using a portable ultrasound device (Logiq-e, GE HealthCare, Boston, MA, USA) with a 9 L linear probe (12 MHz).

SECONDARY OUTCOMES:
Blood biomarkers of kynurenine pathway metabolites | Baseline and 12 weeks
  Plasma levels of KP metabolites [tryptophan (TRP), kynurenine (KYN), quinolinic acid (QUINA), and kynurenic acid (KYNA)], will be measured using commercially available Enzyme-Linked Immunosorbent Assay (ELISA) kits.
Blood biomarkers of inflammation | Baseline and 12 weeks
  Pro-inflammatory cytokines [interleukin-6 (IL-6), tumor necrosis factor-alpha (TNF-α), and interferon-gamma (IFN-y)] will be measured using commercially available Enzyme-Linked Immunosorbent Assay (ELISA) kits.
Blood biomarkers of endothelial injury | Baseline and 12 weeks
  Plasma levels of soluble P-selectin, vascular cell adhesion molecule-1 (sVCAM-1), and intercellular adhesion molecule-1 (sICAM-1) will be assessed using the Human Cardiovascular Disease Panel 2 magnetic kit (EMD Millipore Corporation, MA, USA), with a sensitivity greater than 0.079 ng/ml.
Vascular function | Baseline and 12 weeks
  Endothelial-dependent and -independent vascular function will be assessed by venous occlusion plethysmography
Maximal oxygen consumption | Baseline and 12 weeks
  Maximal oxygen consumption will be collected breath-by-breath using a silicone mask (Hans Rudolph®, Shawnee, USA) connected to an Ultima CardiO2 metabolic cart (Medical Graphics®, Saint Louis, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Borges, PhD, Principal Investigator — Rio de Janeiro State University
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
Unnamed data collected and research results will be stored in a cloud-based system (Dropbox) and may be accessed after permission granted by the principal investigator.

REFERENCES:
- [Derived] Paz GA, Rangel MV, Farias CL, Soares ALC, Langner E, Teixeira T, Dutra PML, Bouskela E, Farinatti P, Souza MDGC, Borges JP. Acute and chronic effects of physical exercise on atherosclerosis, kynurenine pathway, endothelial function and inflammation in patients with coronary artery disease: a clinical trial protocol. BMJ Open Sport Exerc Med. 2025 Feb 10;11(1):e002432. doi: 10.1136/bmjsem-2024-002432. eCollection 2025. PMID 39944998